CLINICAL TRIAL: NCT01060644
Title: Maxillary Sinus Floor Elevation Following Simultaneous Implant Installation Without Graft Material
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: CMC-08-0015-CTIL
Record Dates: First submitted 2010-01-31; First posted 2010-02-02 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Insufficient Bone Volume in Posterior Maxilla
Keywords: Maxillary Sinus; Bone Augmentation; Dental Implant; Sinus Membrane

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study describes and evaluates the surgical protocol for sinus mucosal lining elevation of the maxillary sinus for Dental Implant Insertion without Bone grafting Underneath the Sinus Membrane.

DETAILED DESCRIPTION:
Restoration of lost dentition in the severely atrophic posterior maxilla has for the last 2 decades been successfully treated with various sinus augmentation techniques and installation of dental implants. The use of graft material is anticipated to be necessary; however, recent studies have demonstrated that the mere lifting of the sinus mucosal lining and simultaneous placement of implants result in bone formation. This study was conducted in order to evaluate simultaneous sinus mucosal lining elevation and installation of dental implants without any graft material.

The present study describes and evaluates a modification of the surgical protocol for sinus mucosal lining elevation and simultaneous installation of osseointegrated implants with a MIS implant system (Seven ™) ,in 20 patients.

Preoperative Examination: (Screening):

1. Medical History
2. Clinical Examination

   1. Oral hygiene.
   2. Oral mucosa condition.
   3. Number of missing teeth in the posterior maxilla.
3. Radiographic Examination (CT and Panoramic X-ray)

   1. Sinus Maxillary condition.
   2. Sub-antral bone height.
   3. Bone jaw condition. Selected patients under the "inclusion criteria" will be included in the study after they will have explanation and signed on informed consent.

Surgery:

All patients will be operated on under local anesthesia (2% Xylocaine Dental with epinephrine 1:100,000;) or General anesthesia ( the type of the anesthesia will be decided by the patients) at Carmel medical center Haifa.. Preoperative antibiotics will orally administered 45 minutes before surgery; patients routinely received 2 g of Augmentin or 600 mg of clindamycin (when allergic to penicillin).and 6mg of Dexamethasone 1 hour before surgery.

Surgical Technique:

The posterior maxillary edentulous area and the maxillary sinus wall will be exposed via a crestal incision and a buccal muco-periosteal flap will be raised. Osteotomy in a oval or rectangular fashion will be made with round Drill 5 mm radius in the anterior wall of the sinus, 5 to 6 mm cranial to the intended implant site (Fig 1). With small sharp elevators the cortical bony window will be pulled in the sinus cavity.

Perforations of various sizes of the sinus mucosal lining will be treated by drilling small holes in the bone above the cortical window to elevate and suture the mucosal lining to that level using absorbable sutures (Vicryl 6-0). If there is success in this technique we will use a small piece of periosteum (taken from the buccal flap) which will be placed as a lid over a perforation of the sinus mucosal lining. If the perforations are so small (less than 1 mm) then further dissection of the mucosal lining and "tenting" by the implants will be considered satisfactory for a blood clot to form around the implants.

After the elevation, implants will be installed in the residual sub-antral bone. The remaining bone height will be recorded with a depth gauge during surgery. Primary implant stability will be noted manually at installation. A stabilizing wrench will be used when removing the implant carrier in all cases.

To achieve implant stability in the cases of small remaining levels of vertical subantral bone, the protocol of installing the MIS system dental implant was modified in its last preparation step. The final conical burr was leveled into the bone 1 to 2 mm less than the recommended standard protocol in cases with only 2 to 3 mm residual bone. Thus, a slightly smaller hole for the implant was prepared and the implant could be placed with better primary stability, utilizing the effect of the conical design and the retention of the microthreads in the superior part, adding an extra effect to the placement and thereby achieving sufficient primary stability. The compartment around the implants under the sinus mucosal lining in the sinus floor will be filled with blood from surrounding bleeding (Fig 2), and dental membrane (Zimmer Ltd.) will be placed on the open window, then the incision will be closed with resorbable sutures (Vicryl 3/0. Ethicon Inc

Postoperative Care:

Analgesics will be prescribed with Optalgin or with a nonsteroidal anti-inflammatory drug for 1 to 2 weeks following the surgery. Antibiotic treatment will be continue for 10 days postoperatively with Augmentin 875mg Twice a day (or clindamycin, 300 mg 3 times daily for penicillin allergic patients). Patients should be instructed not to blow their nose and to use nasal spray saline for 14 days after surgery. Wearing dentures will not be allowed for 10 days following the surgery.

Patients will be reviewed and sutures taken out after 7 to 10 days. Clinical and Radiological Follow-up The patient will be recalled to the out patient clinic in Carmel Medical Center, for a follow up. All patients will be checked in the surgery site and x-ray radiograph will be made.

Radiological follow up:

Periapical radiographs and Panoramic X-ray will be used for measurements of 1) the height of the residual alveolar bone at each implant site, and 2) the height of newly formed bone in the maxillary sinus in relation to each implant. Measurements will be made manually with a millimeter scale. The cervical micro-threaded area of the implant will be used as a reference point during measurement.

Criteria for considering the procedure as successful:

1. Successful implants ( no pain, no infection, stable implants) at the uncovering procedure.
2. Periapical and panoramic x-ray at the endpoint shows a bone formation around the implant inside the maxillary sinus.

Uncovering of the implant will be done 6 month after the surgery. All patients will be operated on under local anesthesia (2% Xylocaine Dental with epinephrine 1:100,000;) the implant instillation area and the maxillary sinus wall will be exposed via a crestal incision and a buccal mucoperiosteal flap will be raised.

1. A healing cap will be inserted in the implant.
2. A punch of 2mm biopsy will be take from the maxillary wall. The incision will be closed with resorbable sutures (Vicryl 3/0. Ethicon Inc) around the healing cap.

The referring dentists will carried out the prosthetic rehabilitation after two weeks for the uncovering procedure. All patients will be recalled for follow up after the prosthetic rehabilitation 2 and 4 months in our out patients clinic.

Statistics Descriptive statistics will be used and the correlation of results will be confirmed with linear regression analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patient.
2. Patients that have a rehabilitation dentist.
3. Healthy conditions of Maxillary Sinuses and Oral Mucosa.
4. Healthy bone determined by Panoramic X-ray.
5. Sub-antral bone at least 4 mm as measured on CT.
6. Have a good oral hygiene condition.
7. Patient that does not participate in other clinical study.
8. Patient able to read and understand and sign the informed consent.

Exclusion Criteria:

1. Unhealthy patients, with recorded medical history diseases as: diabetes, mellitus, heart diseases, renal failure, osteoporosis.
2. Patients treated with anticoagulation medication (Coumadin, Plavix).
3. Patients treated with Oral Bisphosphonate drugs (as Fosalan).
4. Patient with a history of Chemotherapy or Radiotherapy treatment.
5. Unhealthy conditions of Maxillary Sinuses.
6. Patient without prosthetic rehabilitation treatment plan ) approved by the referred dentist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients (women, men) with a range of a age 18-65 years will be consecutively included. The patients will be referred to the Department of Oral and Maxillofacial Surgery, Carmel Medical Center, Haifa, for dental implant treatment in the posterior maxilla from every Dental Clinic in Israel
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
CT evaluation before Dental Implant uncovering | In the end of the treatment
CT evaluation of bone regeneration | In the end of each treatment

CONTACTS AND LOCATIONS:
Overall Officials: Samer Srouji, DMD, Ph.D, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel